CLINICAL TRIAL: NCT02502682
Title: Effect of Daily Chlorhexidine Bathing on Clostridium Difficile Rates on the General Medical Floor in Patients Receiving Antibiotics
Brief Title: Chlorhexidine Bathing Effect on Clostridium Difficile Rates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jared Brooks (Other)
Collaborators: Northwestern Medicine (Other)
Responsible Party: Sponsor-Investigator, Jared Brooks, Co-Investigator, Northwestern Medicine
Organization: Northwestern Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDiff070115
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Clostridium Difficile
Keywords: Chlorhexidine bathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Receive the bathing standard of care.
- Interventional (Experimental): Receive daily bathing with 2% Chlorhexidine gluconate bathing wipes.
  Interventions: Drug: Sage 2% Chlorhexidine Gluconate Cloth Patient Preoperative Skin Preparation

INTERVENTIONS:
Drug: Sage 2% Chlorhexidine Gluconate Cloth Patient Preoperative Skin Preparation — Daily bathing.
  Arms: Interventional

SUMMARY:
Clostridium difficile (C. diff.) infections, whether nosocomial or community borne, may present with profound diarrhea, especially in those patients receiving antibiotics. Based on a preliminary review of hospital data, the investigators have found that these symptomatic c. diff infections occur with a relatively high incidence at Delnor Hospital. Notwithstanding their high mortality, one recent study attributes a near quadrupling of hospitalization costs to c. diff infections. Chlorhexidine baths have been shown in multiple randomized trials to help reduce the incidence of highly virulent pathogens and hospital acquired infections. Further, several studies show a favorable effect of reducing the incidence of c. diff infections by using Chlorhexidine baths on ICU patients. Far fewer studies, however, have focused on the effects of these baths on general medical/surgical wards. This investigation seeks to study the effect of the daily use of 2% Chlorhexidine gluconate wipes in patients on the general medical/surgical wards who are exposed to antibiotics for a suspected or confirmed infection.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of antibiotics for suspected or confirmed infection.
* Admitted to the 2600 General/Medical ward at Delnor Hospital.

Exclusion Criteria:

* Antibiotics only for surgical prophylaxis
* Not mentally capable
* Cannot provide consent in English
* Pregnant
* Documented chlorhexidine allergy
* Patient is a prisoner
* Health system employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Relative Risk of C-diff infection | up to 12 months
  Study data will cease to be collected after 300 participants have been enrolled or until 12 months have elapsed. Data will be collected and assessed monthly.
Duration of Hospital stays | expected average of six days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Poustinchian, D.O., Principal Investigator — Hospitalist - Northwestern Medicine Regional Medical Group
Locations (1):
- Northwestern Medicine - Delnor Hospital, Geneva, Illinois, United States